CLINICAL TRIAL: NCT05029973
Title: A Study to Evaluate the Efficacy and Safety of the Hepatic Arterial Infusion Chemotherapy(HAIC) Combined With Sintilimab and Bevacizumab Biosimilar in Unresectable Hepatocellular Carcinoma.
Brief Title: HAIC Combined With Sintilimab and Bevacizumab Biosimilar for Unresectable HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAICDD
Record Dates: First submitted 2021-08-29; First posted 2021-09-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sintilimab; Bevacizumab Biosimilar; HAIC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): HAIC Combined With Sintilimab and Bevacizumab Biosimilar
  Interventions: Drug: HAIC; Drug: Sintilimab; Drug: Bevacizumab Biosimilar

INTERVENTIONS:
Drug: HAIC — hepatic arterial infusion (HAI) of oxaliplatin, fluorouracil/leucovorin (FOLFOX) treatment
  Other Names: Hepatic Artery Infusion Chemotherapy; FOLFOX
Drug: Sintilimab — 200mg IV d1,Q3W
  Other Names: IBI308
Drug: Bevacizumab Biosimilar — 7.5mg/kg IV d1,Q3W
  Other Names: IBI305

SUMMARY:
To Evaluate the Efficacy and Safety of the Hepatic Arterial Infusion Chemotherapy(HAIC) Combined With Sintilimab and Bevacizumab Biosimilar in the Treatment of Patients With Unresectable Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent should be signed before implementing any trial-related procedures;
* Age ranges from 18 to 75 years old.
* CNLC-IIb to IIIb HCC based on the Criteria for diagnosis and treatment of hepatocellular carcinoma (2019 edition)

  * At least ≥ 1 measurable lesions per mRECIST;
  * Child-Pugh grade A or B;
  * ECOG PS scores 0-1;
* No prior therapy for HCC.
* Expected survival time > 6 months;
* Sufficient organ functions, the subjects need to meet the following laboratory indicators:

  * No blood transfusion, no use of hematopoietic stimulators (including g-csf, gm-csf, EPO and TPO) and infusion of human albumin preparations within 14 days prior to screening:Neutrophil absolute count ≥1.5×10^9/L;Platelet count ≥ 100×10^9/L;Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN); or total bilirubin > ULN but direct bilirubin ≤ ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 × ULN;
  * Serum creatinine ≤ 1.5 × ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥ 60 ml/min;
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN
  * Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH exceeds the normal range, the subjects can also be included in the group in case total T3 (or FT3) and FT4 are within the normal range;
  * Myocardial enzyme spectrum should be within the normal range (if the investigator comprehensively judges that the simple laboratory abnormality is not clinically significant, the subject is also included);
* Female subjects of childbearing age should receive a urine or serum pregnancy test and the result is negative, 3 days prior to accept the first study drug administration (day 1 of cycle 1). In case the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Meanwhile, voluntary use of appropriate contraceptive methods shall be taken during the observation period and within 8 weeks of the last administration of the study drug; Women of non-bearing age are defined as at least 1 year after menopause, or those who have undergone surgical sterilization or hysterectomy; For males, appropriate contraceptive methods should be taken during the observation period and within 8 weeks after the last dose of the study drug.
* If there is a risk of pregnancy, all subjects (regardless of male and female) need to adopt contraceptives with an annual failure rate of less than 1% during the entire treatment period until 120 days after the last administration of the study drug (or 180 days after the last chemotherapeutic drug administration).

Exclusion Criteria:

* known as Inhibition of fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC；Previous HCC recurrence；Hepatic encephalopathy has been clinically diagnosed in the past 6 months .
* Autoimmune hepatitis (requiring liver puncture).
* History of organ transplantation or hepatic encephalopathy.
* Diffuse hepatoma.
* Clinical symptoms requiring drainage including pleural effusion, ascites, and pericardial effusion.
* History of nephropathy or nephrotic syndrome.
* Bleeding from a varicose vein in the esophagus or gastric fundus caused by portal hypertension in the past 6 months; Presence of severe (G3) varicose veins identified by endoscopy 3 months prior to initial administration; Evidence of portal hypertension (including imaging findings that the length of the spleen exceeds 10 cm and the platelets lower than 100), with a high risk of hemorrhage assessed by the investigator.
* Arteriovenous thromboembolic events in the past 6 months, including history of myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary artery embolism, deep vein thrombosis or any other serious thromboembolism. Implantable venous infusion port or catheter-derived thrombosis, or superficial venous thrombosis, except for those with stable thrombosis after conventional anticoagulation therapy.
* Severe bleeding tendency or coagulation dysfunction, or under thrombolytic therapy.
* Acceptance of preventive use of low-dose low-molecular-weight heparin (such as Enoxaparin 40 mg/day), except for vitamin K antagonists (such as warfarin).
* Requiring long-term medication for the inhibition of platelet function, such as aspirin, dipyridamole or clopidogrel.
* Uncontrollable hypertension, systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg after optimized medical treatment, history of critical hypertension or hypertensive encephalopathy.
* Symptomatic congestive heart failure (New York Heart Association class II-IV), symptomatic or poorly controlled arrhythmia, congenital long QT syndrome history or QTc > 500 ms corrected at screening (calculated using the Fridericia method).
* History of gastrointestinal perforation and or fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection, complicated by chronic diarrhea), Crohns disease, ulcerative colitis, or long-term chronic diarrhea in the past 6 months.
* Received major surgery (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures within 4 weeks prior to the first administration, except for received tissue biopsy or other minor surgery within 7 days prior to the first administration, venipuncture catheterization for intravenous infusion.
* Past and present history of lung diseases including pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severely impaired lung functions.
* Acute or chronic active hepatitis B or C infection.
* Active tuberculosis (TB), under anti-tuberculosis treatment or anti-tuberculosis treatment within 1 year prior to the first administration.
* Infected by human immunodeficiency virus (HIV) and known syphilis infection.
* Severe infections in active phase or poorly controlled clinically. Severe infection within 4 weeks prior to the first administration.
* Have used immunosuppressive drugs within 4 weeks before the first dose
* Received live attenuated vaccines within 4 weeks before the first dose or plan to receive live attenuated vaccines during the study period
* Received Chinese medicine with anti-tumor indications, or received drugs with immunomodulatory effect within 2 weeks before the first administration
* Received any anti-PD-1 antibody, anti-PD-L1/L2 antibody, anti-CTLA4 antibody, or other immunotherapy
* Allergic to Sintilizumab, Bevacizumab preparations and excipients, or had severe allergic reactions to other monoclonal antibodies in the past
* Received treatment from other clinical trials within 4 weeks before the first dose
* Female subjects who are pregnant or breastfeeding
* Other conditions that the subjects are not suitable to participate in this study according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate ( ORR) | Up to 2 years
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  Defined as the time from the date of treatment start to the date of death
Events Free Survival (EFS) | Up to 2 years
  Defined as the time from enrollment to disease progression, recurrence or death (whichever occurs first)
Surgical conversion rate | Up to 2 years
  Defined as the incidence rate of patients that receive surgical resection.
R0 resection rate of patients who accepted surgical resection | Up to 2 years
  Defined as the proportion of patients undergoing radical resection to the total patients accepted surgical resection
Pathological complete response (pCR) rate of patients who accepted surgical resection | Up to 2 years
  Defined as the proportion of patients whose tumor and lymph node completely disappeared to the total patients accepted surgical resection
Adverse Events (AEs) | Up to 2 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0 and complications of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China